CLINICAL TRIAL: NCT03525561
Title: Influences of Acetazolamide on Endurance Exercise Performance and Cognitive Function During Acute Exposure to Hypobaric Hypoxia
Brief Title: Acetazolamide and Exercise Performance at Altitude
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: M-10729
Record Dates: First submitted 2018-03-16; First posted 2018-05-15 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Hypoxia; Exercise Performance; Cognitive Function; Dexterity
MeSH Terms: conditions — Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Subjects will serve as their own controls. Will exercise during simulated altitude exposure twice, once with acetazolamide and once with placebo.
Who Masked: Participant
Masking Description: Single-blind use of acetazolamide where participant is not informed. Goal is to evaluate effect (or lack thereof) on exercise performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- acetazolamide arm (Active Comparator): This is the arm of the study in which the volunteers will take the acetazolamide (Diamox) pill.
  Interventions: Drug: Acetazolamide Pill
- placebo arm (Placebo Comparator): This is the arm of the study in which volunteers will take the placebo.
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Acetazolamide Pill — Subjects will take acetazolamide pill (Diamox), 500 mg/ day, and assess effect on exercise performance during 30-hour exposure to 3,500 m simulated altitude.
  Other Names: Diamox
  Arms: acetazolamide arm
Drug: Placebo pill — Subjects will take placebo pill and then we will assess exercise performance during 30-hour exposure to 3,500 m simulated altitude.
  Arms: placebo arm

SUMMARY:
The goals of the present study are to evaluate whether the most common, and effective, treatment for acute mountain sickness (AMS), acetazolamide (AZ), has a negative, positive, or no influence on exercise performance, cognitive performance, or manual dexterity in young healthy subjects during simulated altitude exposure. AMS represents a serious challenge to the health and performance of the Warfighter who may need to rapidly deploy to high altitude. However, there have been concerns that AZ might alter or impair endurance exercise performance, and possibly fine motor skills. These would represent major limitations to the use of this drug in a Warfighter who has a specific timeframe in which to accomplish mission tasks. In the present project, we will use exposure to simulated altitude in the USARIEM hypobaric chamber to quantify the impact, if any, of AZ on endurance exercise performance following rapid ascent to 3500 meters (m) in unacclimatized lowlander volunteers. The study will be conducted using a randomized, single-blind, placebo-controlled crossover study design. Ten male and female volunteers will complete one orientation day, one VO2peak day, three days of familiarization testing at sea level (SL), then two rounds of experimental testing. Each round of experimental testing consists of six days including four days to establish baseline euhydration, followed by a 30 hour (hr) exposure to 3500 m. Volunteers will have a two week break between experimental testing rounds for washout of any effects of altitude acclimation. During one experimental round, volunteers will take two doses of AZ each day (Phase 1: 250 mg/dose,500 mg/day, Phase 2: 125 mg/dose, 250 mg/day) starting 48 hr prior to their altitude exposure and continuing for the 30 hr stay at high altitude. During the other experimental condition, volunteers will be given a placebo at the same time points as the doses of AZ. Prior to altitude exposure, AMS will be evaluated and volunteers will then ascend to a simulated altitude of 3500 m, where they will remain for 30 hr. Volunteers will rest at altitude for an hr, after which they will complete an AMS questionnaire, resting ventilation measurements, provide a blood sample and complete cognitive and finger dexterity testing. Subjects will then perform 15 minutes (min) of steady state (SS) treadmill exercise at 40-45% of SL VO2peak and a 2 mile treadmill time trial (TT). Volunteers will stay overnight in the hypobaric chamber with research staff supervision. The following morning, metabolic and blood measurements will again be completed, after which volunteers will perform the exercise testing for a second time. Cognitive and finger dexterity testing will be performed before volunteers return to sea level (i.e., "descend" from the simulated altitude). The results of the proposed study will, for the first time, provide quantitative evidence regarding whether AZ treatment impairs endurance exercise performance in the context of a Warfighter-relevant endurance exercise task.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet all of the following criteria to be included in the study:

* Male or female, age 18-45
* In good health as determined by Office of Medical Support and Oversight (OMSO) General Medical Clearance
* Passed his/her most recent Army Physical Fitness Test (APFT; military volunteers only) or exercise at least 2 times per week (civilian volunteers)
* Willing to not exercise, drink alcoholic beverages, or consume caffeinated products for 24 hours before each testing session.
* Willing not to consume carbonated beverages during the experimental phases of the study (this does not include the two week break between experimental phases)
* Willing to stay and sleep in an altitude chamber (the size of a dorm room) ~60 hours total (two ~30 hr exposures).
* Body mass index (BMI) ≤ 28.5

Exclusion Criteria:

* Females who are pregnant or planning to become pregnant during the study
* Taking dietary supplements, prescriptions, or over the counter medication, other than a contraceptive (unless approved by OMSO and PI)
* Born at altitudes greater than 2,100 m (~7,000 feet; Examples include Santa Fe, New Mexico; Laramie, Wyoming; Etc.)
* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas more than 1,200 m for five days or more within the last 2 months (Examples include Ft. Huachuca, Arizona; Lima, Peru; Feldberg, Germany; etc.)
* Physical problems/injuries associated with walking or running on a treadmill
* Allergy to skin adhesive
* Abnormal blood count (For example: hemoglobin (Hb) outside of the normal ranges (Normal [Hb] Males = 12.6-17.7 g/dL; Females = 11.1-15.9 g/dL) or hematocrit (Hct) outside of the normal ranges (Normal Hct Males = 37.5-51.0%; Females = 34.0-46.6%) levels, presence of abnormal blood chemicals (hemoglobin S or sickle cell traits)
* Prior HAPE (high altitude pulmonary edema) or HACE (high altitude cerebral edema) diagnosis
* Smokers or tobacco/nicotine users (unless have quit more than 4 months prior)
* Presence of asthma or respiratory tract infections (unless more than 1 month prior or approved by OMSO).
* Allergy to sulfa drugs (Acetazolamide)
* Evidence of apnea or other sleeping disorders
* History of neurologic (e.g. stroke, seizure), speech, facial muscle disorder or injuries preventing from producing normal range of hand and finger motion
* Experiencing colds, coughs, or sinus infections
* Food allergies/intolerances to gluten and/or dairy
* Low blood Na+/K+ values ( Na+: < 135 mmol/L, K+: <3.5 mmol/L)
* Kidney, liver or adrenal dysfunction
* Breastfeeding mothers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Endurance exercise performance | Exercise performance will be assessed during a 30-hour simulated altitude exposure, once during placebo and once during acetazolamide administration
  the primary outcome measure is performance of a 2-mile treadmill time trial (self-paced) at simulated altitude.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Charkoudian, Ph.D., Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- Natick Soldier Systems Center, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided